CLINICAL TRIAL: NCT01674010
Title: A Prospective, Randomized, Double-Blind, Placebo-Controlled, Phase 2 Safety and Efficacy Study of Oral ELND005 as an Adjunctive Maintenance Treatment in Patients With Bipolar I Disorder
Brief Title: Safety and Efficacy Study of ELND005 as an Adjunctive Maintenance Treatment in Bipolar I Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business Decision
Sponsor: OPKO Health, Inc. (Industry)
Collaborators: Elan Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ELND005-BPD201; 2012-001935-30 (EudraCT Number)
Record Dates: First submitted 2012-08-24; First posted 2012-08-28 (Estimated); Results first posted 2015-10-12 (Estimated); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Bipolar 1 Disorder
MeSH Terms: interventions — scyllitol; Lamotrigine; Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lamotrigine or Valproic acid + ELND005 (Experimental): Lamotrigine or valproic acid plus ELND005 film coated tablets, 500mg BID for up to 48 weeks
  Interventions: Drug: ELND005; Drug: Lamotrigine; Drug: Valproic acid
- Lamotrigine or Valproic acid + placebo (Placebo Comparator): Lamotrigine or valproic acid plus matched placebo BID for up to 48 weeks
  Interventions: Drug: Lamotrigine; Drug: Valproic acid; Drug: Placebo

INTERVENTIONS:
Drug: ELND005
  Other Names: Scyllo-inositol
  Arms: Lamotrigine or Valproic acid + ELND005
Drug: Lamotrigine
Drug: Valproic acid
Drug: Placebo
  Arms: Lamotrigine or Valproic acid + placebo

SUMMARY:
The primary purpose of this study is to determine whether ELND005 is effective in the maintenance treatment of bipolar 1 disorder when added to other therapies.

ELIGIBILITY:
Inclusion Criteria:

* Meets the DSM-IV-TR criteria for BPD I by the SCID, prior to the Screening Visit.
* Has a history in the last 3 years of ≥ 1 manic or mixed episodes of sufficient severity that required hospitalization and/or treatment with a mood stabilizer or antipsychotic, or confirmed by a family member or medical records to ensure the episode fulfills the DSM-IV-TR criteria.
* Has experienced a mood episode of any polarity within 4 months prior to the Screening Visit and responded to StOC therapy.
* Is euthymic at the Screening Visit (ie, score of ≤ 12 on the MADRS and a score of ≤ 12 on the Y-MRS).
* Is receiving maintenance treatment for his or her BPD I with either LTG or VPA; on stable doses for past 4 weeks and therapeutic drug levels (total VPA 50--125 µg/mL and LTG 10-50 µmol/L or as deemed appropriate by the investigator). Dose adjustments made for tolerability reasons will be acceptable.

A study patient must meet the following additional criteria to be eligible for randomization in the Double-blind Randomization Phase of this study:

- Maintained in a stable euthymic state during Phase 1, defined as Y-MRS and MADRS scores of ≤ 12, with the following exceptions: a maximum of 2 nonconsecutive excursions will be allowed throughout Phase 1. Excursions are defined as Y-MRS or MADRS scores >12 but ≤ 16.

Exclusion Criteria:

* Woman of childbearing potential who is unwilling or unable to use an acceptable method of birth control or is using a prohibited contraceptive method.
* Is found to be actively suicidal on the C-SSRS (answer of "yes" to question 4 or 5 [current or over the last 30 days]) or a score of ≥4 on the MADRS item 10 at the Screening Visit.
* Has suboptimally treated thyroid disease as evidenced by thyroid-stimulating hormone (TSH) >3 mIU/L at the Screening Visit.
* Has received electroconvulsive therapy (ECT) during the current episode or within 6 months prior to the Screening Visit.
* Has an estimated glomerular filtration rate <40 mL/min/1.73 m2 according to the Modification of Diet in Renal Disease formula.

A study patient who meets ANY of the above and ANY of the criteria below will not be eligible for enrollment in the Double-blind Randomization Phase of this study:

* Has current signs or symptoms of psychosis.
* Has become actively suicidal as defined by C-SSRS answer of "yes" to question 4 or 5 (current or over the last 30 days) and/or has a score of ≥4 on MADRS item 10.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 309 (Actual)
Dates: Start 2012-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (74):
- United States (39):
  - Elan Investigational Site, Birmingham, Alabama
  - Elan Investigational Site, Glendale, Arizona
  - Elan Investigational Site, Phoenix, Arizona
  - Elan Investigational Site, Little Rock, Arkansas
  - Elan Investigational Site, Cerritos, California
  - Elan Investigational Site, Costa Mesa, California
  - Elan Investigational Site, Escondido, California
  - Elan Investigational Site, Garden Grove, California
  - Elan Investigational Site, National City, California
  - Elan Investigational Site, Oceanside, California
  - Elan Investigational Site, Palo Alto, California
  - Elan Investigational Site, Riverside, California
  - Elan Investigational Site, San Diego, California
  - Elan Investigational Site, Santa Ana, California
  - Elan Investigational Site, Stanford, California
  - Elan Investigational Site, Norwich, Connecticut
  - Elan Investigational Site, North Miami, Florida
  - Elan Investigational Site, Oakland Park, Florida
  - Elan Investigational Site, Tampa, Florida
  - Elan Investigational Site, Atlanta, Georgia
  - Elan Investigational Site, Roswell, Georgia
  - Elan Investigational Site, Creve Coeur, Missouri
  - Elan Investigational Site, St Louis, Missouri
  - Elan Investigational Site, Lincoln, Nebraska
  - Elan Investigational Site, Marlton, New Jersey
  - Elan Investigational Site, Fresh Meadows, New York
  - Elan Investigational Site, New York, New York
  - Elan Investigational Site, Raleigh, North Carolina
  - Elan Investigational Site, Beachwood, Ohio
  - Elan Investigational Site, Cincinnati, Ohio
  - Elan Investigational Site, Cleveland, Ohio
  - Elan Investigational Site, Oklahoma City, Oklahoma
  - Elan Investigational Site, Philadelphia, Pennsylvania
  - Elan Investigational Site, Charleston, South Carolina
  - Elan Investigational Site, Houston, Texas
  - Elan Investigational Site, Hurst, Texas
  - Elan Investigational Site, San Antonio, Texas
  - Elan Investigational Site, Salt Lake City, Utah
  - Elan Investigational Site, Bellevue, Washington
- Bulgaria (5):
  - Elan Investigational Site, Kardzhali
  - Elan Investigational Site, Pazardzhik
  - Elan Investigational Site, Sofia
  - Elan Investigational Site, Varna
  - Elan Investigational Site, Vratsa
- Canada (7):
  - Elan Investigational Site, Edmonton, Alberta
  - Elan Investigational Site, Kelowna, British Columbia
  - Elan Investigational Site, Halifax, Nova Scotia
  - Elan Investigational Site, Chatham, Ontario
  - Elan Investigational Site, Kingston, Ontario
  - Elan Investigational Site, London, Ontario
  - Elan Investigational Site, Toronto, Ontario
- Czechia (2):
  - Elan Investigational Site, Prague
  - Elan Investigational Site, Strakonice
- France (5):
  - Elan Investigational Site, Bully-les-Mines
  - Elan Investigational Site, Dole
  - Elan Investigational Site, Élancourt
  - Elan Investigational Site, Nîmes
  - Elan Investigational Site, Toulouse
- Poland (4):
  - Elan Investigational Site, Bydgoszcz
  - Elan Investigational Site, Gdansk
  - Elan Investigational Site, Lodz
  - Elan Investigational Site, Tuszyn
- Romania (4):
  - Elan Investigational Site, Brasov
  - Elan Investigational Site, Bucharest
  - Elan Investigational Site, Craiova
  - Elan Investigational Site, Sibiu
- Spain (4):
  - Elan Investigational Site, Torrevieja, Alicante
  - Elan Investigational Site, Oviedo, Principality of Asturias
  - Elan Investigational Site, Barcelona
  - Elan Investigational Site, Vitoria-Gasteiz
- Turkey (Türkiye) (4):
  - Elan Investigational Site, Ankara
  - Elan Investigational Site, Diyarbakır
  - Elan Investigational Site, Edirne
  - Elan Investigational Site, Istanbul

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Treatment Phase 1 ELND005 500 mg BID: ELND005 500mg BID for 16 weeks
- Phase 2 Placebo: Double Blind Randomization (Phase 2)
- Phase 2 ELND005 500 mg BID: Randomization Phase 2 ELND005 500 mg BID
Period: Open Treatment Phase 1
Arm/Group | Open Treatment Phase 1 ELND005 500 mg BID | Phase 2 Placebo | Phase 2 ELND005 500 mg BID
Started | 309 | 0 | 0
Completed | 129 | 0 | 0
Not Completed | 180 | 0 | 0
Not completed — Adverse Event | 10 | 0 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Lost to Follow-up | 19 | 0 | 0
Not completed — Physician Decision | 9 | 0 | 0
Not completed — Protocol Violation | 7 | 0 | 0
Not completed — Sponsor Decision | 79 | 0 | 0
Not completed — Did not remain in a stable remission | 30 | 0 | 0
Not completed — Withdrawal by Subject | 25 | 0 | 0
Period: Randomization Phase 2
Arm/Group | Open Treatment Phase 1 ELND005 500 mg BID | Phase 2 Placebo | Phase 2 ELND005 500 mg BID
Started | 0 | 65 | 64
Completed | 0 | 3 | 3
Not Completed | 0 | 62 | 61
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 1 | 2
Not completed — Mood episode recurrence | 0 | 8 | 2
Not completed — Physician Decision | 0 | 0 | 2
Not completed — Pregnancy | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Sponsor Decision | 0 | 42 | 45
Not completed — Withdrawal by Subject | 0 | 8 | 7

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 309
Age, Continuous [Mean (Standard Deviation); unit: years]
  Phase 1(n=309) | 44.3 (11.09)
  Phase 2 Placebo (n=65) | 44.5 (10.65)
  Phase 2 ELND005 500mg BID(n=64) | 44.6 (10.61)
Sex/Gender, Customized [Number; unit: participants]
  Phase 1 Male | 146
  Phase 1 Female | 163
  Phase 2 Placebo Male | 34
  Phase 2 Placebo Female | 31
  Phase 2 ELND005 500 BID Male | 32
  Phase 2 ELND005 500 BID Female | 32
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino Phase 1 | 23
  Hispanic or Latino Phase 2 Placebo | 4
  Hispanic or Latino Phase 2 ELND005 500 BID | 6
  Not Hispanic or Latino Phase 1 | 284
  Not Hispanic or Latino Phase 2 Placebo | 60
  Not Hispanic or Latino Phase 2 ELND005 500 BID | 58
  Unknown Phase 1 | 2
  Unknown Phase 2 Placebo | 1
  Unknown Phase 2 ELND005 500 BID | 0
Region of Enrollment [Number; unit: participants]
  North America | 210
  Europe | 99

OUTCOME MEASURES:

1. Primary Outcome: Treatment Emergent Adverse Events
Description: The study was terminated early so no efficacy analysis was done, safety data are reported.
Time Frame: up to 48 weeks
Population: TEAEs reported for Phase 2 were from the entire study period
Measure: Number; unit: participants
Arm/Group | Open Treatment Phase 1 ELND005 500 mg BID | Phase 2 Placebo | Phase 2 ELND005 500 mg BID
Number analyzed (Participants) | 309 | 65 | 64
participants | 153 | 45 | 45

2. Secondary Outcome: Proportion of Study Participants With Recurrence of Any Mood Episode
Time Frame: up to 48 weeks
Population: Study was prematurely terminated, no data were collected for this Outcome Measure
Arm/Group | Open Treatment Phase 1 ELND005 500 mg BID | Phase 2 Placebo | Phase 2 ELND005 500 mg BID
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Time to Recurrence of a Depressive Episode
Time Frame: up to 48 weeks
Population: Study was prematurely terminated, no data were collected for this Outcome Measure
Arm/Group | Open Treatment Phase 1 ELND005 500 mg BID | Phase 2 Placebo | Phase 2 ELND005 500 mg BID
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Time to Recurrence of a Manic/Hypomanic or a Mixed Episode
Time Frame: up to 48 weeks
Population: Study was prematurely terminated, no data were collected for this Outcome Measure
Arm/Group | Open Treatment Phase 1 ELND005 500 mg BID | Phase 2 Placebo | Phase 2 ELND005 500 mg BID
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were recorded for each patient starting from the time the consent form was signed until the completion of the study.
Arm/Group | Open Treatment Phase 1 ELND005 500 mg BID | Phase 2 Placebo | Phase 2 ELND005 500 mg BID
Serious Adverse Events (participants affected / at risk) | 12/309 | 3/65 | 3/64
Other Adverse Events (participants affected / at risk) | 153/309 | 45/65 | 45/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open Treatment Phase 1 ELND005 500 mg BID (N=309) | Phase 2 Placebo (N=65) | Phase 2 ELND005 500 mg BID (N=64)
Depression (Psychiatric disorders) | 3 | 0 | 0
Bipolar I Disorder (Psychiatric disorders) | 1 | 0 | 0
Cardiac disorder (Cardiac disorders) | 1 | 0 | 0
Embolic stroke (Cardiac disorders) | 1 | 0 | 0
Food Poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 1
Gastroenteritis (Gastrointestinal disorders) | 1 | 0 | 0
Hemolytic anemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Impulsive Behaviour (Psychiatric disorders) | 1 | 0 | 0
Mania (Psychiatric disorders) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
Abortion spontaneous (Reproductive system and breast disorders) | 0 | 1 | 0
Diplopia (Eye disorders) | 0 | 0 | 1
Intentional self-injury (Psychiatric disorders) | 0 | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open Treatment Phase 1 ELND005 500 mg BID (N=309) | Phase 2 Placebo (N=65) | Phase 2 ELND005 500 mg BID (N=64)
Gastrointestinal disorders (Gastrointestinal disorders) | 29 | 12 | 11
General disorders and administration site conditions (General disorders) | 10 | 2 | 5
Infections and infestations (Infections and infestations) | 47 | 20 | 20
Injury poisoning and procedural complications (Injury, poisoning and procedural complications) | 19 | 15 | 11
Investigations (Investigations) | 13 | 8 | 8
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 9 | 2 | 5
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 18 | 11 | 10
Nervous system disorders (Nervous system disorders) | 35 | 13 | 11
Psychiatric disorders (Psychiatric disorders) | 63 | 15 | 13
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 4
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 12 | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days